CLINICAL TRIAL: NCT01320280
Title: Single-arm, Open-label, Single-center Phase II Study Evaluating the Efficacy and Safety of BIBW 2992 (Afatinib) for the Treatment of Patients With HER2-positive, Hormone-refractory Prostate Cancer After Failure of Treatment With Docetaxel or Ineligible for Treatment With Docetaxel
Brief Title: BIBW 2992 (Afatinib) for the Treatment of Patients With HER2-positive, Hormone-refractory Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: unexpectedly slow recruitment
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.138
Record Dates: First submitted 2011-03-17; First posted 2011-03-22 (Estimated); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Refractory Cancer
Keywords: Prostate cancer, BIBW 2992 (Afatinib) , HER inhibitor
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIBW 2992 (Afatinib) (Experimental): BIBW 2992 (Afatinib) 50mg daily continuously (oral medication)
  Interventions: Drug: BIBW 2992 (Afatinib)

INTERVENTIONS:
Drug: BIBW 2992 (Afatinib) — 50 mg BIBW 2992 (Afatinib) tablets daily continuously

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, BIBW 2992 (Afatinib) has on patients and their advanced prostate cancer which does not respond to hormone or chemotherapy any more. Only patients with tumors which have an increased amounts of a protein called HER2 on their cell surface will be included.

BIBW 2992 (Afatinib) is a drug which in advanced clinical testing in lung and breast cancer.

DETAILED DESCRIPTION:
This is a phase II study of BIBW 2992 (Afatinib) in patients with hormone and chemotherapy (docetaxel) refractory, HER2 overexpressing prostate cancer. The exploratory study following a two stage Gehan design. In the first stage 29 patients with be treated. Additional patients will be recruited in a second stage depending on the number of responding patients in the first step. Patients will receive BIBW 2992 (Afatinib) orally at a dose of 50 mg daily. Response to therapy will be scored according to PSA values (Bubley criteria) and to CT scans (RECIST criteria). Patients will be seen at 2 or 4 weeks intervals by a medical professional while on the medication for toxicity assessment and physical examination. Disease evaluations will occur at baseline and every 2 months thereafter. These evaluations will include PSA testing and CT Scans (if appropriate).

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent
* Age ≥ 18 years
* Patients must have histological proven, hormone-refractory prostate cancer
* Patients must have failed prior therapy with docetaxel or must be ineligible for treatment with docetaxel
* Patients must have ECOG performance status ≤ 2
* Patients must not have received any prior therapy targeting EGFR or HER2
* Patients must have adequate bone marrow, renal and hepatic function
* Patients must not have a history of severe heart disease
* Patients must not have had a myocardial infarction within the previous six months
* Patients must have normal left ventricular ejection fraction (LVEF ≥ normal limit of institution)
* Patients must not have symptomatic brain or leptomeningeal metastatic disease
* Patients must have recovered from previous treatment-related adverse effects to National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (CTCAE) grade ≤ 1

Exclusion Criteria:

* Prior treatment with EGFR/HER2-targeted small molecules or antibodies, i.e. trastuzumab and/or lapatinib
* Known pre-existing interstitial lung disease
* Radiotherapy, chemotherapy, hormone therapy (with the exception of GnRH agonists), immunotherapy or surgery (other than biopsy) within 4 weeks prior to start of treatment with BIBW2992. GnRH-agonists are allowed at the discretion of the investigator.
* Active brain metastases (defined as stable for < 4 weeks and/or symptomatic and/or requiring changes of treatment with anticonvulsants or steroids within the past 4 weeks and/or leptomeningeal disease). Patients with known history of brain metastases should undergo a baseline brain image to ensure that the disease is stable.
* Any other current malignancy or malignancy diagnosed within the past five (5) years (other than non-melanomatous skin cancer).
* Significant or recent acute gastrointestinal disorders with diarrhoea as a major symptom, e.g. Crohn's disease, malabsorption or CTC grade ≥ 2 diarrhoea of any aetiology.
* History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of 3, unstable angina or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to randomisation.
* Cardiac left ventricular function with resting ejection fraction of less than 50%.
* Any other concomitant serious illness or organ system dysfunction which in the opinion of the investigator would either compromise patient's safety or interfere with the evaluation of the safety of the test drug.
* Absolute neutrophil count (ANC) < 1500 / mm³.
* Platelet count < 75,000 / mm³
* Calculated creatinine clearance < 60 ml / min (using Cockcroft-Gault formula for GFR estimate) or serum creatinine > 1.5 times upper limit of normal.
* Uncontrolled hypercalcemia
* Patients unable to comply with the protocol.
* Known hepatitis B infection, known hepatitis C infection or known HIV carrier.
* Known or suspected active drug or alcohol abuse.
* Requirement for treatment with any of the prohibited concomitant medications
* Any contraindications for therapy with BIBW 2992.
* Known hypersensitivity to BIBW 2992.
* Use of any investigational drug within 4 weeks of start of treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Objective PSA responses according to Bubley criteria | every two months
  Bubley criteria see Bubley GJ, et al. Eligibility and response guidelines for phase II clinical trials in androgen-independent prostate cancer: recommendations from the Prostate-Specific Antigen Working Group. J Clin Oncol 1999; 17: 3461-3467

SECONDARY OUTCOMES:
Objective response rate (ORR) based on Response Evaluation Criteria in Solid Tumours (RECIST 1.1) | every 2 months
Duration of PSA-response (Bubley criteria) or objective responses | every 2 months
Safety | every 4 weeks
  Description AEs according to CTC criteria

CONTACTS AND LOCATIONS:
Overall Officials: Walter Fiedler, M.D:, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Background] Yap TA, Vidal L, Adam J, Stephens P, Spicer J, Shaw H, Ang J, Temple G, Bell S, Shahidi M, Uttenreuther-Fischer M, Stopfer P, Futreal A, Calvert H, de Bono JS, Plummer R. Phase I trial of the irreversible EGFR and HER2 kinase inhibitor BIBW 2992 in patients with advanced solid tumors. J Clin Oncol. 2010 Sep 1;28(25):3965-72. doi: 10.1200/JCO.2009.26.7278. Epub 2010 Aug 2. PMID 20679611
- [Result] Minner S, Jessen B, Stiedenroth L, Burandt E, Kollermann J, Mirlacher M, Erbersdobler A, Eichelberg C, Fisch M, Brummendorf TH, Bokemeyer C, Simon R, Steuber T, Graefen M, Huland H, Sauter G, Schlomm T. Low level HER2 overexpression is associated with rapid tumor cell proliferation and poor prognosis in prostate cancer. Clin Cancer Res. 2010 Mar 1;16(5):1553-60. doi: 10.1158/1078-0432.CCR-09-2546. Epub 2010 Feb 23. PMID 20179235